CLINICAL TRIAL: NCT00512967
Title: The Inflammatory and Antioxidant Status in Pulmonary Sarcoidosis, Idiopathic Pulmonary Fibrosis and COPD: a Potential Role for Antioxidants
Brief Title: The Occurence of Inflammation and Oxidative Stress in Lung Diseases
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Dr. A.W. Boots, Maastricht University
Other Study IDs: MEC 03-112
Record Dates: First submitted 2007-07-19; First posted 2007-08-08 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2008-02

CONDITIONS: Interstitial Lung Diseases; Sarcoidosis; Idiopathic Pulmonary Fibrosis; COPD
Keywords: oxidative stress; antioxidants; inflammation; quercetin
MeSH Terms: conditions — Lung Diseases, Interstitial; Sarcoidosis; Idiopathic Pulmonary Fibrosis; Pulmonary Disease, Chronic Obstructive; Inflammation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood samples were collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- sarcoidosis: 21 onset patients, non-treated
- IPF: 15 IPF patients, partially treated
- COPD: 15 COPD patients within 24 hours after their last exacerbation
- controls: 25 healthy controls, matched for age and gender

SUMMARY:
Reactive oxygen species (ROS) are suggested to play a pivotal role in ILD. Little is known, however, about the endogenous antioxidant levels in ILD that can offer protection against ROS. It is expected that the high amount of ROS present in ILD will reduce the antioxidant levels. Therefore, antioxidant therapy to strengthen this reduced antioxidant defense might be efficacious in ILD treatment. Since ROS are capable of initiating and mediating inflammation, antioxidant therapy might also mitigate elevated inflammation. A candidate for antioxidant therapy is the flavonoid quercetin that is known for its anti-oxidative and anti-inflammatory capacities.

The aim of the present study is to determine the antioxidant and inflammatory status in ILD, i.e. sarcoidosis and idiopathic pulmonary fibrosis (IPF). Furthermore, to evaluate the possible anti-inflammatory effects of antioxidants, the effect of quercetin will be examined on the ex vivo LPS-induced cytokine production in ILD

DETAILED DESCRIPTION:
Interstitial lung diseases (ILD) include various chronic lung disorders such as sarcoidosis and idiopathic lung fibrosis (IPF). In the Netherlands the incidence of sarcoidosis is approximately 20-25 per 100.000 inhabitants whereas that of IPF is approximately 1000-1500 new cases each year.

In short, three different stages in the development of ILD can be discerned. Firstly, the lung tissue is damaged. In sarcoidosis this damage is thought to be antigen-driven, multisystemically and leading to the formation of granuloma. Moreover, it is suggested that genetic factors play an important role in the genesis of sarcoidosis. In IPF the exact etiology of this damage is unknown, but it has been speculated to be inflicted by an unidentified stimulus that produces repeated episodes of acute lung injury Secondly, the walls of the air sacs in the lung become inflamed as a reaction to the caused damage. This results in the activation of inflammatory cells like macrophages that cause the expression of pro-inflammatory cytokines, especially interleukin-10 and tumour necrosis factor (TNF)-alpha, in the lungs.

Finally, scarring (or fibrosis) begins in the interstitium (or tissue between the air sacs) and the lung becomes stiff, causing an irreversible loss of the tissue's ability to transfer oxygen.

It is well-known that inflammation plays a key-role in the occurrence and progression of ILD, although the long-lasting hypothesis that inflammation alone leads to fibrosis is being questioned at the moment. Conventional treatment of ILD comprises nonspecific anti-inflammatory agents such as glucocorticoids (prednisone) and other immune-suppressing medication such as cyclophosphamide, methotrexate and gamma-interferon. However, all these therapies fail to be completely efficacious, suggesting that inflammation alone is indeed not solely responsible for the occurrence and progression of ILD. Paradoxically, anti-TNF-α agents such as infliximab and thalidomide have recently shown some beneficial effects in sarcoidosis.

A pivotal role for reactive oxygen species (ROS) in all three stages has also been proposed. Various biomarkers of oxidative stress, i.e. exhaled ethane and both 8-isoprostane and oxidized proteins in the bronchoalveolar fluid, are elevated in ILD patients of different clinical stages. However, only little is known about the effect of this elevated oxidative stress on the endogenous antioxidant levels present in ILD. Interestingly, clinical administration of an antioxidant, i.e. N-acetylcysteine (NAC), to IPF patients has recently demonstrated that this slows the deterioration of vital capacity and carbon monoxide diffusing capacity (DLCO) at 12 months. This supports the hypothesis that oxidative stress is involved in ILD and proofs the principle of antioxidant treatment in ILD.

It is well-known that oxidative stress and inflammation are intertwined and that the pro-inflammatory cytokine TNF-alpha is capable of stimulating oxidative stress in various cells and tissues. As a result, the preliminary beneficial effects of anti-TNF-alpha agents combined with the preliminary beneficial effects of antioxidants in ILD may indicate that a new strategy of treatment of ILD should ideally combine the reduction of both the oxidative stress and the inflammation occurring in these diseases.

Recently, much attention has been given to the potential health-beneficial properties of flavonoids, natural occurring polyphenolic compounds, and to quercetin, the most commonly occurring flavonoid, in particular. Quercetin is known to be a powerful antioxidant and to possess some anti-inflammatory effects. It is therefore tempting to speculate that quercetin could exert positive effects in ILD.

Since the anti-oxidative and inflammatory changes in ILD are still not exactly known, the aim of the present study is to determine both the anti-oxidant and the inflammatory status in ILD, i.e. sarcoidosis and fibrosis. Furthermore, the possible anti-inflammatory effect of antioxidants on LPS-induced cytokine production, exemplified with the flavonoid quercetin, will be examined.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of pulmonary sarcoidosis, IPF or COPD
* no treatment for sarcoidosis
* last exacerbation not more than 24 hours ago for COPD
* healthy controls
* no smoking for sarcoidosis and IPF

Exclusion Criteria:

* pregnancy
* use of vitamins or food supplements
* clinical diagnosis (and treatment) of other diseases
* symptoms of sarcoidosis in other organs besides the lung

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: lung patients visiting the out-patient clinic of the Academic Hospital Maastricht
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2005-09; Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aalt Bast, PhD, Study Chair — Maastricht University; Agnes W Boots, PhD, Principal Investigator — Maastricht University; Guido R Haenen, PhD, Study Director — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands